CLINICAL TRIAL: NCT05053776
Title: Clinical and Laboratory Predictors of Respiratory Morbidities in Children With Cerebral Palsy at Assiut University Children Hospital
Brief Title: Clinical and Laboratory Predictors of Respiratory Morbidities in CP Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Remonda Ramsis Hennis (Other)
Responsible Party: Sponsor-Investigator, Remonda Ramsis Hennis, Resident doctor at pediatrics department, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Respiratory morbidities in CP
Record Dates: First submitted 2021-03-25; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Relationship between respiratory morbidities and cerebral palsy in children

DETAILED DESCRIPTION:
Identification of symptoms,signs,severity and outcomes of respiratory morbidities in children with Cp

ELIGIBILITY:
Inclusion Criteria:

* children with CP from 1 month to 18 years

Exclusion Criteria:

* neonates with Cp CP patients more than 18 years old

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Identification of different respiratory problems in children with cerebral palsy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Chest auscultation | Baseline
  Identify any respiratory abnormalities in CP patients

SECONDARY OUTCOMES:
Chest X-ray | Baseline
  Identify any chest infection in CP patients